CLINICAL TRIAL: NCT05872958
Title: A Phase I, Randomized, Safety and Pharmacokinetics Study of AZD3152 in Healthy Adults (Little DIPPER)
Brief Title: Dose Exploration Intramuscular/Intravenous Prophylaxis Pharmacokinetic Exposure Response Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: D7000C00004
Record Dates: First submitted 2023-05-15; First posted 2023-05-24 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: COVID-19
Keywords: Coronavirus disease 2019 (COVID-19); Prophylaxis setting
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- AZD3152 Dose X (IM) (Experimental): Participants will receive dose X of AZD3152 on Day 1 as a single IM injection.
  Interventions: Drug: AZD3152
- AZD3152 Dose X (IV) (Experimental): Participants will receive dose X of AZD3152 on Day 1 as an IV infusion.
  Interventions: Drug: AZD3152
- AZD3152 Dose Y (IM) (Experimental): Participants will receive dose Y of AZD3152 on Day 1 as 2 sequential IM injections.
  Interventions: Drug: AZD3152
- AZD3152 Dose Y (IV) (Experimental): Participants will receive dose Y of AZD3152 on Day 1 as an IV infusion.
  Interventions: Drug: AZD3152
- AZD3152 Dose Z (IV) (Experimental): Participants will receive dose Z of AZD3152 on Day 1 as an IV infusion.
  Interventions: Drug: AZD3152
- Pooled placebo (Placebo Comparator): Participant will receive placebo on Day 1 either via IM injection or IV infusion.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: AZD3152 — AZD3152 will be administered via IM injection or IV infusion, as per the assigned arms.
  Arms: AZD3152 Dose X (IM); AZD3152 Dose X (IV); AZD3152 Dose Y (IM); AZD3152 Dose Y (IV); AZD3152 Dose Z (IV)
Other: Placebo — Placebo is a matching volume of 0.9% sodium chloride, will be administered via IM injection or IV infusion, as per the assigned arms.
  Arms: Pooled placebo

SUMMARY:
This is a dose exploration study to evaluate the safety and pharmacokinetics (PK) of AZD3152 in healthy adult male and female participants, across different dose levels and routes of administration (ie, Intramuscular [IM] injection and Intravenous [IV] infusion).

DETAILED DESCRIPTION:
The study will be conducted in the United States of America.

Eligible healthy participants will be randomized to receive either AZD3152 or placebo administered IM or IV, across 5 fixed-dose cohorts. Participants will receive a single dose of AZD3152/placebo.

Cohort 1: Dose X of AZD3152 or placebo, as an IM injection Cohort 2: Dose X of AZD3152 or placebo, administered IV Cohort 3: Dose Y of AZD3152 or placebo, as an IM injection Cohort 4: Dose Y of AZD3152 or placebo, administered IV Cohort 5: Dose Z of AZD3152 or placebo, administered IV

The study will comprise of:

* A Screening Period of maximum 28 days.
* A Treatment Period of one Day.
* A Follow-up Period of 12 months after study intervention (Day 365).

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female participants.
* Participants have suitable veins for cannulation or repeated venipuncture.
* Negative SARS-CoV-2 RT-PCR or SARS-CoV-2 rapid antigen test result at Visit 1.
* Body weight ≥ 45 kg and ≤ 110 kg and body mass index ≥ 18 and <32 kg/m2 at Screening.
* Able to complete the Follow-up Period up to Day 365 as required by the protocol.

Exclusion Criteria:

* History of any clinically important disease or disorder.
* Receipt of any immunoglobulin (either COVID-19 or non-COVID related) or blood products within 6 months prior to Day 1.
* Receipt of an EVUSHELD monoclonal antibody (mAb) against SARS-CoV-2 within last 15 months before Day 1.
* Receipt of a COVID-19 vaccine within 14 days prior to Visit 1.
* SARS-CoV-2 infection within one month prior to Visit 1 (confirmed either by laboratory testing or a rapid test [including at-home testing]).
* Women who are pregnant, lactating, or of childbearing potential and not using a highly effective method of contraception or abstinence from at least 4 weeks prior to study intervention administration and until at least 6 months after study intervention administration.
* Known or suspected congenital or acquired immunodeficiency, or receipt of immunosuppressive therapy,
* Any clinically important illness, medical/surgical procedure, or trauma within 4 weeks of the first administration of study intervention. This includes any acute (time-limited) or febrile (temperature ≥ 38.0°C [100.4ºF]) illness/infection on day prior to or day of planned dosing; participants excluded for transient acute illness may be dosed if illness resolves within the Screening Period or may be rescreened once.
* Any abnormal laboratory values as described in protocol.
* Any known HIV or hepatitis B or C infection at Screening.
* History of alcohol or substance abuse that in the opinion of the Investigator might interfere with the trial conduct or completion.
* Known hypersensitivity to AZD3152.
* Previous hypersensitivity or severe adverse reaction following administration of a mAb.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 98 (Actual)
Dates: Start 2023-05-19 (Actual); Primary Completion 2024-08-20 (Actual); Study Completion 2024-08-20 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse event | Until Day 91
  Evaluation of the safety of IM or IV administration of AZD3152 will be done.
Number of participants with serious adverse event | Until Day 365 or early discontinuation visit (EDV [approximately 19 months])
  Evaluation of the safety of IM or IV administration of AZD3152 will be done.
Number of participants with adverse event of special interest | Until Day 365 or EDV (approximately 19 months)
  Evaluation of the safety of IM or IV administration of AZD3152 will be done.
Serum concentration of AZD3152 | Pre-dose, and Day 1 until Day 365 or EDV (approximately 19 months)
  Pharmacokinetics (PK) characterization of AZD3152 in serum after a single IM or IV dose.
Maximum observed concentration (Cmax) of AZD3152 | Pre-dose, and Day 1 until Day 365 or EDV (approximately 19 months)
  PK (Cmax) characterization of AZD3152 in serum after a single IM or IV dose.
Time to reach maximum observed concentration (tmax) of AZD3152 | Pre-dose, and Day 1 until Day 365 or EDV (approximately 19 months)
  PK (tmax) characterization of AZD3152 in serum after a single IM or IV dose.
Terminal elimination half-life (t1/2) of AZD3152 | Pre-dose, and Day 1 until Day 365 or EDV (approximately 19 months)
  PK (t1/2) characterization of AZD3152 in serum after a single IM or IV dose.
Area under the serum concentration-curve from 0 to the last quantifiable concentration (AUClast) of AZD3152 | Pre-dose, and Day 1 until Day 365 or EDV (approximately 19 months)
  PK (AUClast) characterization of AZD3152 in serum after a single IM or IV dose.
Area under concentration-time curve from 0 to infinity (AUCinf) of AZD3152 | Pre-dose, and Day 1 until Day 365 or EDV (approximately 19 months)
  PK (AUCinf) characterization of AZD3152 in serum after a single IM or IV dose.
Apparent total body clearance (CL/F) of AZD3152 (IM administration only) | Pre-dose, and Day 1 until Day 365 or EDV (approximately 19 months)
  PK (CL/F) characterization of AZD3152 in serum after a single IM.
Apparent volume of distribution based on terminal phase (Vz/F) of AZD3152 (IM administration only) | Pre-dose, and Day 1 until Day 365 or EDV (approximately 19 months)
  PK (Vz/F) characterization of AZD3152 in serum after a single IM.
Total body clearance (CL) of AZD3152 (IV administration only) | Pre-dose, and Day 1 until Day 365 or EDV (approximately 19 months)
  PK (CL) characterization of AZD3152 in serum after a single IV.
Volume of distribution based on terminal phase (Vz) of AZD3152 (IV administration only) | Pre-dose, and Day 1 until Day 365 or EDV (approximately 19 months)
  PK (Vz) characterization of AZD3152 in serum after a single IV.
Volume of distribution at steady state (Vss) of AZD3152 (IV administration only) | Pre-dose, and Day 1 until Day 365 or EDV (approximately 19 months)
  PK (Vss) characterization of AZD3152 in serum after a single IV.

SECONDARY OUTCOMES:
Number of participants with anti-drug antibody (ADA) to AZD3152 | Pre-dose, Days 15, 31, 91, 181, and Day 365
  Evaluation of ADA responses to AZD3152.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Research Site, Anniston, Alabama
  - Research Site, Cullman, Alabama
  - Research Site, Scottsdale, Arizona
  - Research Site, Orlando, Florida

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All requests will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: Redated CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D7000C00004&attachmentIdentifier=c9dd1921-ccae-4a5c-87fa-56ea2ea8714f&fileName=D7000C00004-Redacted_CSR_Synopsis.pdf&versionIdentifier=
- See also: Results of this clinical trial are available on www.astrazenecaclinicaltrials.com — http://astrazenecagrouptrials.pharmacm.com/ST/Submission/Search